CLINICAL TRIAL: NCT00740805
Title: A Phase I Study of ABT-888 in Combination With Cyclophosphamide in Solid Tumors or Non-Hodgkin Lymphoma
Brief Title: Veliparib, Cyclophosphamide, and Doxorubicin Hydrochloride in Treating Patients With Metastatic or Unresectable Solid Tumors or Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00262; NCI-2009-00262 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000600234; 050803; 050803 (Other: Rutgers Cancer Institute of New Jersey); 7998 (Other: CTEP); P30CA072720 (NIH); U01CA132194 (NIH); U01CA099118 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-08

CONDITIONS: Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma; Solid Neoplasm
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (veliparib, cyclophosphamide, doxorubicin) (Experimental): GROUP I: Patients receive veliparib PO every 12 hours on days 1-4 and cyclophosphamide IV over 60 minutes on day 3.
  GROUP II: Patients receive veliparib PO every 12 hours on days 1-4, cyclophosphamide IV over 60 minutes on day 3, and doxorubicin hydrochloride IV over 15 minutes on day 3.
  GROUP III: Patients receive veliparib PO every 12 hours on days 1-7, cyclophosphamide IV over 60 minutes on day 1, and doxorubicin hydrochloride IV over 15 minutes on day 1.
  GROUP IV: Patients receive veliparib PO every 12 hours on days 1-14, cyclophosphamide IV over 60 minutes on day 1, and doxorubicin hydrochloride over 15 minutes on day 1.
  In all groups, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib, cyclophosphamide, and doxorubicin hydrochloride when given together in treating patients solid tumors or non-Hodgkin lymphoma that has spread to other areas of the body or cannot be removed by surgery. Veliparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and doxorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib, cyclophosphamide, and doxorubicin hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the maximally tolerated dose (MTD) and dose limiting toxicity (DLT) of cyclophosphamide when combined with escalating doses of ABT-888 (veliparib).

II. Identify the maximally tolerated dose (MTD) and dose limiting toxicity (DLT) of cyclophosphamide and doxorubicin (doxorubicin hydrochloride) when combined with escalating doses of ABT-888.

SECONDARY OBJECTIVES:

I. Evaluate any effect of ABT-888 on the systemic clearance of parent cyclophosphamide and the dose normalized area under the curve (AUC) of 4-hydroxy (4-OH) cyclophosphamide when used in combination, using historical single-agent cyclophosphamide and 4-OH data.

II. Evaluate any effect of cyclophosphamide administration on the systemic pharmacokinetics of ABT-888 and its primary metabolite A-925088 (M8), by comparing pharmacokinetic (PK) parameters of ABT-888 on day 1 (before cyclophosphamide) and day 3 (with cyclophosphamide administration); PK samples for analysis will not be collected from patients enrolled after 2/15/2012.

III. Evaluate inhibition of poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) using an immunoassay designed to measure PAR levels in baseline and on-study peripheral blood mononuclear cells (PBMC) samples; PBMC samples for PAR analysis will not be collected from patients enrolled after 2/15/2012.

IV. Evaluate gamma H2A histone family, member X (H2AX) at baseline and on-study circulating tumor cell samples to evaluate the point of maximal deoxyribonucleic acid (DNA) damage from the combination of cyclophosphamide and doxorubicin with ABT-888.

OUTLINE: This is a dose-escalation study of veliparib and cyclophosphamide.

GROUP I: Patients receive veliparib orally (PO) every 12 hours on days 1-4 and cyclophosphamide intravenously (IV) over 60 minutes on day 3.

GROUP II: Patients receive veliparib PO every 12 hours on days 1-4, cyclophosphamide IV over 60 minutes on day 3, and doxorubicin hydrochloride IV over 15 minutes on day 3.

GROUP III: Patients receive veliparib PO every 12 hours on days 1-7, cyclophosphamide IV over 60 minutes on day 1, and doxorubicin hydrochloride IV over 15 minutes on day 1.

GROUP IV: Patients receive veliparib PO every 12 hours on days 1-14, cyclophosphamide IV over 60 minutes on day 1, and doxorubicin hydrochloride over 15 minutes on day 1.

In all groups, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patients with either solid tumors or non-Hodgkin's lymphoma are eligible

  * At the recommended Phase II dose level, an additional 6 to 12 patients in each group with the following criteria will be enrolled: documented breast cancer (BRCA)1/BRC2 mutation, triple-negative breast cancer defined as estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and human epidermal growth factor receptor (HER)2-negative, or patients who would benefit from a cyclophosphamide-based regimen
  * On the schedule of ABT-888 given for 7 or 14 days, only patients with metastatic breast cancer will be enrolled
* Patients must be >= 4 weeks since prior chemotherapy or radiation therapy (>= 6 weeks if the last regimen included carmustine [BCNU] or mitomycin C); patients previously treated with cyclophosphamide should not be necessarily excluded
* Patients with non-Hodgkin's lymphoma that is amenable to hematopoietic stem cell transplantation with curative intent may participate only if stem cell transplant is refused or is not indicated
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 2 months
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN), =< 5 x ULN if known hepatic metastases
* Creatinine within normal institutional limits OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.2 X institutional ULN
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients enrolled in a group where the treatment is adriamycin and cycloblastin (AC): ejection fraction >= 50% by multigated acquisition scan (MUGA) or echocardiogram
* Patients must sign informed consent

Exclusion Criteria:

* Concurrent administration of any other investigational agent(s)
* Prior high-dose therapy requiring hematopoietic stem cell transplantation
* Prior anti-cancer treatments involving radioactive pharmaceuticals
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 and/or cyclophosphamide
* Patients receiving any medications or substances that are strong inhibitors or strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP 3A4), cytochrome P450, family 2, subfamily B, polypeptide 6 (2B6), cytochrome P450, family 2, subfamily C, polypeptide 9 (2C9) or cytochrome P450, family 2, subfamily C, polypeptide 19 (2C19) are prohibited; at the time of screening, if the patient is currently receiving any of the listed prohibited medication(s), the medication(s) must be discontinued for a period of no less than 7 days prior to administration of the first dose of study medication in order for the patient to meet study eligibility except for the following substance where the washout should be 6 months: amiodarone
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; New York Heart Association (NYHA) grade II or greater congestive heart failure
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated; NOTE: HIV seropositive patients not receiving combination antiretroviral therapy who have cluster of differentiation (CD)4 cells >= 350/mm^3, no opportunistic infections and meet all eligibility criteria may participate in this study
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain ABT-888 capsules
* Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption (e.g., inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, active peptic ulcer disease) are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* Patients with active central nervous system (CNS) metastases are excluded

  * Patients with CNS metastases that have been treated must be off steroid treatment for > 3 months, be asymptomatic and off steroid treatment prior to study enrollment
  * Patients that have symptoms to suggest CNS metastases should have a brain magnetic resonance imaging (MRI) within 28 days of enrollment to confirm the absence of CNS metastases; contrast computed tomography (CT) is acceptable for patients who are unable to undergo a brain MRI
* Patients with active seizure or a history of active seizure
* Any other medical, social, or psychological condition that may significantly affect safety and/or compliance
* Patients enrolled in a group where treatment is AC: prior doxorubicin exposure of > 300 mg/m^2 or equivalent anthracycline exposure (i.e., epirubicin dose > 540 mg/m^2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-08-18 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
MTD, defined as the dose level that no more than 2/6 or 1/3 patients experience DLT and at least 2/3 or 3/6 patients treated with next higher dose level will have had DLT | 21 days
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0

SECONDARY OUTCOMES:
Change in pharmacokinetic parameters | Day 1, course 1 to day 1, course 2
  A two way analysis of variance model will be used to compare the PK parameters.
Change in gammaH2AX levels (quantification of the time point of maximal DNA damage) | Baseline to up to day 14

CONTACTS AND LOCATIONS:
Overall Officials: Mark N Stein, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States